CLINICAL TRIAL: NCT02329431
Title: Padres Efectivos (Parent Activation): Skills Latina Mothers Use to Get Healthcare for Their Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: University of North Carolina, Greensboro (Other)
Responsible Party: Principal Investigator, Kathleen Thomas, PhD, Fellow and Adjunt Associate Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 13-2106
Record Dates: First submitted 2014-12-29; First posted 2014-12-31 (Estimated); Results first posted 2017-07-07 (Actual); Last update posted 2017-07-07 (Actual); Status verified 2017-04

CONDITIONS: Mental Disorders
Keywords: child mental health, mental health services, Latino families
MeSH Terms: conditions — Mental Disorders | interventions — Self-Help Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- activation curriculum (Experimental): Psycho-social curriculum teaching activation skills
  Interventions: Behavioral: activation curriculum
- support group (Active Comparator): Parent-directed support group
  Interventions: Behavioral: support group

INTERVENTIONS:
Behavioral: activation curriculum — psychosocial activation curriculum
  Arms: activation curriculum
Behavioral: support group — parent directed support group
  Arms: support group

SUMMARY:
The goal of this study is to develop an intervention to teach activation skills to Latino parents who bring children for mental health services.

DETAILED DESCRIPTION:
Background:

Latinos are the largest and fastest growing minority population in the US; by 2050, 2 in 5 children will be Latino. Latino children are disproportionately affected by poverty and other factors associated with increased risk of psychiatric disorder. However, Latino children with mental health needs are half as likely to use services as children in white non-Latino families. Latino families are more likely to report problems getting services, lack of a usual source of care and a medical home, and dissatisfaction with the care they receive. Unmet mental health needs, in turn, are associated with poor outcomes over the lifespan, both economic and social. Assessing the comparative effectiveness of interventions to overcome these disparities is a major national health priority central to PCORI's mission and mandate.

Activation is a promising focus of research to eliminate disparities because it reflects a set of attitudes and skills that people can use to reduce disparities. Our work provides evidence that activation in Latino adults is associated with better quality health care and outcomes; and in African American parents with greater child mental health service use. There is need for further research on parent-focused interventions founded on culturally meaningful concepts to address these needs and disparities.

Objectives:

The long-term goal of this research is to improve the mental health care and outcomes of Latino children with mental health needs. The proposed study will examine the comparative effectiveness of an activation intervention for Latino families raising children with mental health needs by means of three aims:

Aim 1. To identify parent-reported facilitators of Latino child mental health service use amenable to change through parental activation Aim 2. To test the comparative effectiveness of an adapted psycho-educational intervention to teach activation skills adapted for Latino mothers of children with mental health needs compared to a parent support group control Aim 3. To enhance the intervention, based on parent input and lessons learned from the first trial, and test its comparative effectiveness with a parent support group control

Methods:

Qualitative and quantitative data from Latino mothers who have a child with mental health needs (n=294) will be used in a difference-in-difference mixed effects approach to address these aims.

Projected Patient Outcomes:

The proposed study will provide evidence of the comparative effectiveness of an enhanced, culturally sensitive, advocacy skills intervention to build activation among Latino families and improve service use of their children with mental health needs compared to a preliminary adaptation of an existing intervention and to a usual care discussion group. Activation skills are a promising strategy to improve child mental health service use and to bridge cultural differences and disparities with wide-ranging impacts consistent with PCORI's research agenda.

ELIGIBILITY:
Inclusion Criteria:

* For children:

  * seeking services at target clinic
  * maximum age 22 years
* For caregivers:

  * Latino ethnicity
  * bringing child for services to target clinic
  * able to attend a weekly class for 4 weeks
  * able to give informed consent

Exclusion Criteria:

* For children:

  * not living with potential participant caregiver
* For caregiver:

  * not living with target child
  * evidence of emergency mental health needs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2013-08; Primary Completion 2016-07 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen C Thomas, PhD, Principal Investigator — UNC Chapel Hill
Locations (1):
- UNC Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was from a Spanish-language mental health clinic, November 2013 through August, 2015
Pre-assignment Details: Evaluation criteria were focal child not living with potential participant and evidence of urgent parent mental health needs
Period: Overall Study
Arm/Group | Activation Curriculum | Support Group
Started | 92 | 89
Baseline Interview | 87 | 85
Completed | 72 | 76
Not Completed | 20 | 13
Not completed — Lost to Follow-up | 20 | 13

BASELINE CHARACTERISTICS:
Population: Completed a baseline interview
Groups:
- Total: Total of all reporting groups
Arm/Group | Activation Curriculum | Support Group | Total
Number analyzed (Participants) | 87 | 85 | 172
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.3 (6.9) | 36.4 (6.3) | 35.8 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 84 | 168
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 87 | 85 | 172
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 87 | 85 | 172
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 87 | 85 | 172
Medicaid coverage [Count of Participants; unit: Participants] — Target child covered by Medicaid
  Participants | 62 | 62 | 124

OUTCOME MEASURES:

1. Primary Outcome: Patient Activation Measure
Description: The Patient Activation Measure (PAM) captured parent activation on behalf of their child. The PAM is an adult self-report 13-item scale with 4-level Likert responses and scores ranging from 0 to 100. Higher scores indicate higher activation. It is valid with excellent reliability. The PAM has been translated into Spanish and has been used successfully in Latina/o patient and general populations (mean=40). The PAM has also been used to measure activation of parents on behalf of their children (mean=70). A change of 4 points in the PAM is associated with improved health behaviors in the general population.
Time Frame: 1 and 3 months
Population: Completed a baseline interview
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Activation Curriculum | Support Group
Number analyzed (Participants) | 87 | 85
scores on a scale
  patient activation measure 1-month | 88.08 (12.13) | 84.73 (12.65)
  patient activation measure 3-months | 92.75 (10.52) | 91.63 (11.13)

2. Secondary Outcome: 8-item Patient Health Questionnaire (PHQ-8)
Description: Parent depression was measured with the 8-item Patient Health Questionnaire (PHQ-8). The PHQ-8 is scored on a scale from 0 to 27; a higher score reflects greater severity of depression. It has excellent validity and reliability. The parent PHQ-9 has been translated into Spanish and used successfully in Latina/o populations. A change of 5 points in the PHQ-8 is associated with a shift in level of depression.
Time Frame: 1 and 3 months
Population: Completed a baseline interview
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Activation Curriculum | Support Group
Number analyzed (Participants) | 87 | 85
scores on a scale
  patient health questionnaire-8 1-month | 4.63 (5.91) | 3.49 (4.34)
  patient health questionnaire-8 3-months | 3.89 (4.63) | 3.47 (4.43)

3. Secondary Outcome: Parental Stress Scale
Description: Parent stress was measured with the 17-item Parental Stress Scale. The Parental Stress Scale is scored on a scale from 0 to 75, where higher scores reflect greater stress. It has been translated into Spanish, and has been shown to have excellent validity and reliability (for women, mean=22).
Time Frame: 1 and 3 months
Population: Completed a baseline interview
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Activation Curriculum | Support Group
Number analyzed (Participants) | 87 | 85
scores on a scale
  parental stress scale 1-month | 28.51 (7.63) | 29.97 (6.90)
  parental stress scale 3-months | 26.68 (6.69) | 27.25 (6.61)

4. Secondary Outcome: Parent Activation, Qualitative
Description: We collected qualitative data on parent-provider communication after completion of the 4-week MePrEPA (metas, preguntar, escuchar, preguntar para aclarar/goals, questioning, listening, questioning to clarify) and parent support groups, in an effort to capture observed activation. We coded when the parent disagreed with therapist and when the parent mentioned speaking with child's teacher.
Time Frame: 1 month
Population: Completed baseline interview and had an audio-recorded visit
Measure: Count of Participants; unit: Participants
Arm/Group | Activation Curriculum | Support Group
Number analyzed (Participants) | 55 | 63
Participants
  parent disagreed with therapist | 4 | 5
  parent mentioned speaking with child's teacher | 16 | 16

5. Secondary Outcome: Number of Clinic Visits Child Attended Over 4 Months
Description: We collected child attendance at clinic visits during a 4-month window of time, during the 3-month period parents were participating in the study and one additional month following. Child clinic visit attendance was measured by number of visits attended.
Time Frame: baseline to 4-month follow-up
Population: Target child with any scheduled clinic visits
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Activation Curriculum | Support Group
Number analyzed (Participants) | 87 | 84
visits | 4.2 (2.8) | 4.0 (2.8)

6. Secondary Outcome: Child Visit No-shows Over 4 Months
Description: We collected child attendance at clinic visits during a 4-month window of time, during the 3-month period parents were participating in the study and one additional month following. Child clinic visit no-shows were measured by number of visits missed.
Time Frame: baseline to 4-month follow-up
Population: Target child with any scheduled visits
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Activation Curriculum | Support Group
Number analyzed (Participants) | 87 | 84
visits | 0.7 (0.9) | 0.6 (1.0)

ADVERSE EVENTS:
Arm/Group | Activation Curriculum | Support Group
Serious Adverse Events (participants affected / at risk) | 0/92 | 0/89
Other Adverse Events (participants affected / at risk) | 0/92 | 0/89

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No